CLINICAL TRIAL: NCT00561860
Title: Use of a Remote-Monitoring System to Diagnose and Treat Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Philips Respironics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: H06-70411; C06-0411
Record Dates: First submitted 2007-11-19; First posted 2007-11-21 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-03

CONDITIONS: Obstructive Sleep Apnea-hypopnea
Keywords: Obstructive sleep apnea-hypopnea; Telemedicine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): This pathway represents our standard clinical protocol when a patient has been diagnosed with sleep apnea and CPAP therapy is initiated. After prescription of CPAP, all patients will be seen by our CPAP coordinator and oriented to the device during a 20 minute session. Patients are also provided the telephone number of the CPAP coordinator who can be contacted if any problems or questions arise.
- 2 (Experimental): Telemedicine involves the provision or support of direct clinical care via the application of electronic and communicating technology, including the remote monitoring of health status. By providing patient data early in the course of CPAP prescription, we believe that this technology would be immensely useful in improving compliance and acceptance of the device in patients with sleep apnea.
  Interventions: Device: Telemedicine Arm

INTERVENTIONS:
Device: Telemedicine Arm — Telemedicine involves the provision or support of direct clinical care via the application of electronic and communicating technology, including the remote monitoring of health status. By providing patient data early in the course of CPAP prescription, we believe that this technology would be immensely useful in improving compliance and acceptance of the device in patients with sleep apnea.
  Arms: 2

SUMMARY:
Although continuous positive airway pressure (CPAP) is an effective therapy for obstructive sleep apnea-hypopnea (OSAH), one of the major impediments to its use is poor compliance. Adherence with CPAP ranges from 50% to 75%, and subjective reports underestimate actual use. The primary objectives are to determine whether a remote monitoring system improves 3 month compliance (average hours of use/night), and reduces the costs of caring for patients with OSAH who are prescribed CPAP.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether a telemedicine monitoring system can improve the care of patients with OSAH. This system allows close monitoring of patients after prescription of CPAP, and will transmit clinically useful physiologic information (i.e., residual sleep apnea, mask leak, applied pressure, compliance with therapy) daily to the patient's healthcare provider. This should allow early detection of problems with appropriate interventions thereby improving early experience with CPAP, reducing the number of patients who discontinue CPAP therapy and improving overall compliance.

The primary objectives are to determine whether a telemedicine system:1)improves 3 month compliance (average hours of use/night), and 2)reduces the costs of caring for patients with moderate to severe OSAH who are prescribed CPAP.

Secondary objectives are to determine whether this system will improve a variety of other outcomes including: 1) CPAP acceptance (proportion of patients who agree to use CPAP), 2) proportion of high CPAP users (>4 hours average per night), 3) subjective sleepiness, 4) satisfaction with CPAP, 5) side effects with CPAP, 6) # changes in therapy, and 7) time to adequate treatment. In addition, the overall satisfaction of this system will also be assessed.

Telemedicine involves the provision or support of direct clinical care via the application of electronic and communicating technology, including the remote monitoring of health status. By providing patient data early in the course of CPAP prescription, we believe that this technology would be immensely useful in improving compliance and acceptance of the device in patients with sleep apnea.

We intend to perform a randomized controlled trial of this system versus standard care in patients with moderate to severe OSAH. Patients will be randomized to either the 'standard care' arm or the 'telemedicine' arm. To minimize allocation bias, randomization will be performed using sequential numbered envelopes.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for a sleep study to rule out sleep apnea at the Sleep Disorders Program, University of British Columbia. All patients with documented moderate to severe OSAH (AHI≥15 events per hour by PSG) who are prescribed CPAP by their regular sleep physician, and who are willing to accept a trial of CPAP would potentially eligible for the trial.
* Patients must also provide a telephone number that would allow contact during regular office hours if necessary. Patients must also have access to a telephone line in their bedroom that can be used to transmit data with the modem.
* We have decided to only study patients with moderate to severe disease, as these are the patients who are most at risk of future CV disease and motor vehicle crashes. As such, we believe that improving CPAP compliance in this group of patients would be especially important.

Exclusion Criteria:

Patients will be excluded from participating if they:

* Are unable/unwilling to provide informed consent
* Have active cardiopulmonary or psychiatric disease
* Have previously been treated for OSA, or
* Do not reside in the greater Vancouver area.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2007-11; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
CPAP compliance (3 months) and overall cost of patient care | 3 months

SECONDARY OUTCOMES:
CPAP acceptance (proportion of patients who agree to use CPAP), proportion of high CPAP users (>4 hours average per night), subjective sleepiness, satisfaction with CPAP, side effects with CPAP, # changes in therapy, and time to adequate treatment. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Najib Ayas, MD, MPH, Principal Investigator — University of British Columbia; Lisa Cortes, RT, Study Director — University of British Columbia; John Fleetham, MD, Study Director — University of British Columbia
Locations (1):
- Sleep Disorders Program, UBC Hospital, Vancouver, British Columbia, Canada